CLINICAL TRIAL: NCT07185750
Title: Investigation of Biopsychosocial Characteristics According to Catastrophizing of Pain Reported by Parents in Patients Diagnosed With JIA
Brief Title: Investigation of Catastrophizing of Pain Reported by Parents in JIA Patients
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 25/530
Record Dates: First submitted 2025-09-13; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Idiopathic Arthritis (JIA); Childhood Rheumatic Diseases
Keywords: Pain catastrophizing; chronic pain
MeSH Terms: conditions — Arthritis, Juvenile; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases diagnosed with JIA: JIA patients and their parents who visited the rheumatology outpatient clinic of a university hospital. A questionnaire will be administered to the child cases and their parents.
  Interventions: Other: Questionnaire application for JIA cases and their parents

INTERVENTIONS:
Other: Questionnaire application for JIA cases and their parents — Scales will be applied to cases diagnosed with JIA and their parents

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the primary rheumatic disease reported to affect the pediatric population. Research suggests that parents' thoughts and feelings about their child's pain, specifically with JIA diagnosis, may influence treatment compliance. Considering that this situation may also affect children's adherence to treatment, the identification and management of parents' catastrophizing of pain is emphasized as important in improving treatment outcomes. This study aimed to examine the biopsychosocial characteristics of parents of children diagnosed with JIA according to their reported catastrophizing of pain.

ELIGIBILITY:
Inclusion Criteria:

* Between 7-18 years of age
* Diagnosed with JIA
* Individuals who volunteer to participate in the study will be included.

Exclusion Criteria:

* Having advanced heart/lung/liver/kidney disease, neurological disease, or malignancies
* Having undergone major orthopedic surgery
* Not volunteering to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale-Parent (PCS-P) | Baseline
  It is assessed using a 5-point Likert scale ranging from 0 (never) to 4 (always) and consists of 13 items. Similar to the child questionnaire, it assesses 3 domains: rumination, magnification, and helplessness. A total score between 0 and 52 is obtained; higher scores reflect a higher level of catastrophizing in parents.
Pain Catastrophizing Scale-Children (PCS-C) | Baseline
  Consists of 13 items that describe the different thoughts and feelings children may experience when they feel pain. The questionnaire measures three domains: rumination, magnification, and helplessness. All items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (always). Higher scores indicate more catastrophic pain beliefs. The total score ranges from 0 to 52.

SECONDARY OUTCOMES:
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Patient | Baseline
  It is a patient/parent-centered measurement method that helps assess the patient's biopsychosocial aspects, such as disease activity, posture, functional and psychosocial status, fatigue, and school performance. The results from the questions are used to assess the functional status of children, while their psychosocial status is recorded based on their answers to 21 questions (ranging from 0 to 358). A high score indicates a poor psychosocial status.
Childhood Health Assessment Questionnaire (CHAQ) | Baseline
  The CHAQ assesses the functional abilities of children diagnosed with rheumatic diseases in their daily living activities. It consists of eight subscales (dressing and personal care, standing up, eating, walking, body care, reaching, grasping, activities) (0-3) and also assesses pain and general well-being using a visual analog scale (0-100). A high score indicates low functionality.
Juvenile Arthritis Quality of Life Questionnaire (JAQQ) | Baseline
  It consists of 74 items covering various health domains, including physical functioning, emotional well-being, and general symptoms. The items are divided into four dimensions related to the child's quality of life: gross motor function (GMF), fine motor function (FMF), psychosocial function (PF), and systemic or general symptoms (SGS). Each domain is scored on a Likert-type scale from 1 to 7; higher scores indicate poorer health-related quality of life. There is also a "not applicable to me" option for the items. The scale also includes a pain measurement (10 cm Visual Analog Scale (VAS)) to assess pain, but this score is not included in the total score.
Juvenile Arthritis Biopsychosocial Scale-JAB-Q-Family | Baseline
  JAB-Q is a multidimensional questionnaire and a parent (family) form. Developed in Turkish by Ünal and colleagues, the questionnaire is completed by one of the child's parents. The family form evaluates the parents' biopsychosocial status from their own perspective and provides scores ranging from 0 to 102. Higher scores indicate a worse biopsychosocial status.
Child and Adolescent Scale of Participation (CASP) | Baseline
  This is a 20-question survey that evaluates the community participation of children and adolescents in school, neighborhood, and local settings. The survey is divided into four sections: 6 questions about home participation, four questions on neighborhood and community involvement, five questions regarding school participation, and five questions on home and community engagement. It is rated on a scale of "expected for their age (full participation), somewhat limited, very limited, unable to participate, and inapplicable." The survey is completed by the child's family or primary caregiver. The person filling out the questionnaire is asked to select the answer that best describes the child's level of participation. The assessment is scored out of 100 points, with higher scores reflecting a greater level of participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No